CLINICAL TRIAL: NCT04479332
Title: The Change of Critical Patient Managements and Subsequent Influences Under Epidemic of Coronavirus Disease 19 (COVID-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202005094RIND
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2020-07

CONDITIONS: Corona Virus Infection; Critical Illness
Keywords: Coronavirus disease 19 (COVID-19); Critical care; Endotracheal intubation; Cardiopulmonary resuscitation; Stress; Environment contamination
MeSH Terms: conditions — Coronavirus Infections; Critical Illness; COVID-19 | interventions — Intubation, Intratracheal; Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resuscitation Area (Experimental): Critical patient is assigned to the resuscitation area for treatment under medical staff on personal protective equipment; Manpower distribution during tracheal intubation: 1-2 licensed physicians, 2-3 nurses (1 for preparing intubation materials and acts as the assist, 1-2 for administering medications and documentation); Manpower distribution during cardiopulmonary resuscitation: 2 licensed physicians (1 inside resuscitation area, 1 at nurses' station), 4 nurses (2 inside resuscitation area, 2 at the sterile area)
  Interventions: Procedure: Tracheal intubation and cardiopulmonary resuscitation
- Negative Pressure Isolation Room (Experimental): Critical patient is assigned to the negative pressure isolation room for treatment under medical staff on personal protective equipment; Manpower distribution during tracheal intubation: 1 licensed physician, 2 nurses (1 for preparing intubation materials, acts as the assist, and for administering medications; 1 for documentation at the anteroom); Manpower distribution during cardiopulmonary resuscitation: 2 licensed physicians (1 inside negative pressure isolation room, 1 at nurses' station), 5 nurses (2 inside negative pressure isolation room, 1 at the anteroom, 2 at the sterile area)
  Interventions: Procedure: Tracheal intubation and cardiopulmonary resuscitation

INTERVENTIONS:
Procedure: Tracheal intubation and cardiopulmonary resuscitation — Critical patients at the emergency room who require tracheal intubation and/or cardiopulmonary resuscitation will be sequentially allocated to either the resuscitation area or negative pressure isolation room for treatment by the designated medical staff wearing personal protective equipment.

SUMMARY:
In the ER of National Taiwan University Hospital, the critical patients are treated (including tracheal intubation and cardiopulmonary resuscitation) in either resuscitation area or negative pressure isolation rooms based on the past history and present illness. During COVID-19 epidemic, whether sequential changes in environmental and personal protective equipment would change the difference of treatment efficacy and patient safety remains unclear. Whether treating patients in resuscitation area or negative pressure isolation room would cause different physical and psychological stress of medical staff and environmental contamination is also unknown. This study aims to conduct a prospective sequential allocation clinical trial to investigate the success rate, patient safety, physical and psychological stress of medical staff, and the risk of environmental contamination of tracheal intubation and cardiopulmonary resuscitation between the resuscitation area and negative pressure isolation room. The results of the study may be used to improve the protocol and protective policy in treating critical patients during an epidemic.

DETAILED DESCRIPTION:
The critical care of patients with an emergency has always been the clinical challenge to the medical staff in the emergency room (ER). The emergency includes sudden cardiac arrest, respiratory failure, acute conscious change, cardiovascular emergency, sepsis, etc. How to treat these patients appropriately and immediately is an important issue, which may change the disease process and prognosis, and save the life.

Owing to the epidemic of coronavirus disease 19 (COVID-19), several changes in the environmental and personal protective equipment have been made in the ER when treating critical patients. The doctor and nurses need to wear individual protective equipment including Level C protective clothing, goggles, N95 mask, surgical mask, guard panel, hair cap, and double-layered gloves to prevent infectious droplet during tracheal intubation. However, the protective equipment may limit the movement and obstruct the vision and thus result in response delays, difficult intubation, and prolong hand-off period during cardiopulmonary resuscitation. On the other hand, wearing N95 mask, surgical mask and guard panel may impair the communication. Additionally, the medical staff may not have enough time to wear the protective equipment during emergency events, and therefore suffer from a higher risk of infection, which may consequently cause a certain level of psychological stress.

This study aims to conduct a prospective sequential allocation clinical trial to investigate the success rate, patient safety, physical and psychological stress of medical staff, and the risk of environmental contamination of tracheal intubation and cardiopulmonary resuscitation between the resuscitation area and negative pressure isolation room. The results of the study may be used to improve the protocol and protective policy in treating critical patients during an epidemic.

ELIGIBILITY:
Inclusion Criteria for Critical Care Patients:

* showing respiratory distress
* require airway protection
* EOC notified of an out-of-hospital cardiac arrest

Exclusion Criteria for Critical Care Patients:

* age less than 20 years old
* pregnant
* in-hospital cardiac arrest in patients prior to intubation
* confirmed cases of covid-19 prior to intubation
* patient or patient's family refuses the procedure

Inclusion Criteria for Medical Staff:

* staff who attended index intubation or resuscitation are encouraged to answer the survey form

Exclusion Criteria for Medical Staff:

* none

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
The success rate of tracheal intubation between resuscitation area and negative pressure isolation rooms | 6 months
  Comparison between the duration and number of tries needed to intubate a patient, or achieve ROSC in patients requiring cardiopulmonary resuscitation, in resuscitation area and negative pressure isolation rooms.
The patient prognosis between resuscitation area and negative pressure isolation rooms | 6 months
  Comparison between the survival rate of patients who were intubated in the resuscitation area and negative pressure isolation rooms, taking into account the duration of hospital stay, respiratory status (successful extubation, post tracheostomy, etc), and neurological state (using the Glasgow coma score, cerebral performance categories, and overall performance categories) upon discharge from the hospital.
The physical and psychological stress of medical staff | 14 days
  The medical staff involved in the intubation and/or cardiopulmonary resuscitation procedures will be asked to voluntarily fill up a survey form to determine their level of psychological stress. They will also be followed up within 14 days post exposure for covid-19 symptoms and undergo testing and quarantine if needed.
The amount of environmental contamination between resuscitation area and negative pressure isolation rooms | 14 days
  The facilities in both resuscitation area and negative pressure isolation rooms will be sampled and compared for the presence of the coronavirus after each intubation or cardiopulmonary resuscitation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Shan Tsai, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin CH, Lin HY, Wu SN, Tseng WP, Chen WT, Tien YT, Wu CY, Huang CH, Tsai MS. Using a telemedicine-assisted airway model to improve the communication and teamwork of tracheal intubation during the coronavirus disease 2019 pandemic. J Telemed Telecare. 2024 Aug;30(7):1140-1148. doi: 10.1177/1357633X221124175. Epub 2022 Sep 6. PMID 36066025